CLINICAL TRIAL: NCT07007962
Title: A Multi-center, Open-label, Single-arm Study to Evaluate the Efficacy and Safety of Oral Rilzabrutinib in Adults With Immune Thrombocytopenia (ITP) Who Failed First-line Treatment
Brief Title: Study to Evaluate the Efficacy and Safety of Oral Rilzabrutinib in Adults With Immune Thrombocytopenia (ITP) Who Failed First-line Treatment
Acronym: LUNA 4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS18573; U1111-1320-4669 (Registry Identifier: WHO ICTRP)
Record Dates: First submitted 2025-05-20; First posted 2025-06-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rilzabrutinib (Experimental): 400 mg BID
  Interventions: Drug: rilzabrutinib

INTERVENTIONS:
Drug: rilzabrutinib — Pharmaceutical form:Tablet-Route of administration:Oral
  Other Names: SAR444671

SUMMARY:
This is a multinational, open label, single arm study that will evaluate the impact of early multi-immune modulation with rilzabrutinib in adult ITP patients who failed first-line treatment. The study includes a screening period (up to 8 weeks), a primary analysis period (up to 28 weeks), a long-term extension period for selected participants (28 weeks) and a 24-week follow-up period only for eligible participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female participants aged 18 years and older with primary ITP
* Participant received at least a first line therapy and had a history of response while on treatment
* Participant has loss of response, relapse or steroid dependency

Key Exclusion Criteria:

* Participants with Secondary ITP
* Participants with Evans syndrome or history of myelodysplastic syndrome
* Participants with history of lymphoma, leukemia, or any malignancy within the past 5 years except for non-melanoma skin malignancy.
* Participants with history of solid organ transplant
* Participants with history of coagulation or bleeding disorders other than ITP
* Participant received advanced therapy for ITP or was splenectomized
* Pregnancy or nursing The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2027-11-05 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Durable platelet response | Until Week 28
  Defined as the percentage of participants able to achieve platelet counts ≥50 000/μL (or ≥30 000/μL and <50 000/μL and at least double from baseline) for ≥50% of 6 biweekly scheduled platelet measurements and at least 4 non-missing, biweekly visits during the last 12 weeks of the primary analysis period (PAP) in absence of rescue therapy

SECONDARY OUTCOMES:
Overall platelet response | Until Week 28
  Percentage of participants able to achieve 2 platelet counts at least 5 days apart of ≥50 000/μL (or ≥30 000/μL and <50 000/μL and at least double from baseline) without rescue medication in the 4 weeks prior to the first elevated platelet count
Duration of platelet response | Until Week 28
  Cumulative number and proportion of non-missing weeks with platelet counts ≥50 000/μL (or ≥30 000/μL and <50 000/μL and at least double from baseline) in absence of rescue medication in the 4 weeks prior to the elevated platelet count in participants who achieve a response (single platelet count)
Change from baseline in the immune thrombocytopenia bleeding scale (IBLS) score at the end of week 28 | Until Week 28
Percentage of participants able to discontinue or reduce CS dose by 50% or to <5 mg from baseline at the end of week 28 | Until Week 28
Frequency and severity of treatment emergent adverse events (TEAEs, including serious adverse events [SAEs], bleeding TEAEs, adverse event of special interest [AESI] and adverse events leading to discontinuation) | Until Week 80
Percentage of participants with potential clinical significant abnormal (PCSA) | Until Week 80
  PCSA in physical examination, ECG, vital signs, and clinical laboratory test results: serum chemistry and hematology (except for platelet counts included in the primary efficacy endpoint)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - New York Oncology Hematology_Investigational Site Number: 8400010, Albany, New York
  - Community Cancer Trials of Utah_Investigational Site Number: 8400002, Ogden, Utah
- France (3):
  - Investigational Site Number : 2500001, Dijon
  - Investigational Site Number : 2500002, Pessac
  - Investigational Site Number : 2500004, Toulouse
- Investigational Site Number : 6160003, Skorzewo, Poland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS18573 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26780&tenant=MT_SNY_9011